CLINICAL TRIAL: NCT01112618
Title: Pergoveris Non Interventional Study
Brief Title: A Non-interventional Study to Identify the Patients With Severe Luteinizing Hormone Deficiency in the Daily Practice
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: W. Bilger, Merck Serono GmbH, Darmstadt, Germany
Other Study IDs: 200061-500
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2011-04

CONDITIONS: Infertility
Keywords: Infertility; Reproductive technologies, Assisted; r-hFSH; r-hLH; Pergoveris
MeSH Terms: conditions — Infertility; Helping Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This non-interventional study is planned to identify the subjects with severe luteinizing hormone (LH) deficiency in the daily practice. The results will be used for the "Periodic Safety Update Report", which is to be regularly sent to the European Medicines Agency (EMEA) and the responsible German Higher Federal Authority (BfArM).

DETAILED DESCRIPTION:
Female subjects with distinctive follicle stimulating hormone (FSH) and LH deficiency require both FSH and LH. Until now these subjects were treated either with a combination of two recombinant preparations (r-hFSH and r-hLH) or else with a menotropin preparation, composed of urinary human FSH (u-hFSH) and human chorionic gonadotropin (hCG) as LH-replacement.

In Pergoveris™ for the first time both hormones FSH and LH are available as recombinant produced hormones in a combination preparation.

Pergoveris has both hormones i.e. FSH and LH available as recombinant produced hormones in a combination preparation in the ratio 2:1. This study is planned to record data for the stimulation not only in case of the ovarian stimulation with intercourse for the optimum (VZO) but also the intrauterine insemination (IUI) and the ovarian stimulation for the assisted reproduction [in-vitro fertilisation (IVF) and intracytoplasmatic sperm injection (ICSI)] in subjects with severe FSH and LH deficiency and learn more about this subject group and the applied stimulation plan.

Apart from the demographic data, anamnestic details e.g. reason for the infertility, duration of the unfulfilled wish for children, past medical treatment for conception and accompanying illnesses will be documented. The duration of the stimulation with Pergoveris as well as the dose per day will be recorded from the cycle documentations. Follicle sizes and hormones will be documented in accordance with the respectively carried out cycle monitoring. The result of the treatment is related to the number of cycles with ovulation stimulation using hCG, the number of the cycles with puncture, the number of the cycles with embryo transfer, the number and quality of the ova and embryos, on occurred pregnancies and documented abortions. Multiple pregnancies and births will also be recorded.

OBJECTIVES

* To find the reason for the diagnosis of the severe LH deficiency such as e.g. low endogenous LH, amenorrhea, low endometrial thickness or low estradiol level.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects undergoing stimulation with Pergoveris for the ovarian stimulation with VZO or with IUI or in preparation for a technology of the assisted conception such as IVF or ICSI

Exclusion Criteria:

* Subjects receiving combination cycles with clomifen, follitropin beta, urinary FSH, urinary human menopausal gonadotropin (hMG)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing stimulation with Pergoveris for the ovarian stimulation with intercourse for the optimum (VZO) or with IUI or in preparation for a technology of the assisted conception such as IVF or ICSI.
Sampling Method: Probability Sample
Enrollment: 3247 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Reason for diagnosis of severe LH deficiency | 6 months
  The reasons for the diagnosis of severe LH deficiency could be low endogenous LH, amenorrhea, low endometrial thickness, low estradiol levels.

SECONDARY OUTCOMES:
Dose on the first day and the last day of treatment; duration of the stimulation; and the total dose of Pergoveris. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sigbert Jahn, PhD, Study Director — Merck Serono GmbH, Germany
Locations (1):
- Fertility Center Berlin, Spandauer Damm 130, Berlin, Germany

REFERENCES:
- [Derived] Buhler K, Naether OG, Bilger W. A large, multicentre, observational, post-marketing surveillance study of the 2:1 formulation of follitropin alfa and lutropin alfa in routine clinical practice for assisted reproductive technology. Reprod Biol Endocrinol. 2014 Jan 14;12:6. doi: 10.1186/1477-7827-12-6. PMID 24423045